CLINICAL TRIAL: NCT00444340
Title: An Open-Label Multicentre Long-Term Extension Study of Etanercept in Ankylosing Spondylitis
Brief Title: An Open-Label Multicentre Long-Term Extension Study of Etanercept for Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A3-101615
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel (Etanercept)

SUMMARY:
This study is an extension trial of 0881A3-312-EU and is designed to provide information on the safety and efficacy of etanercept in patients with ankylosing spondylitis for up to 3 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Completed study 0881A3-312-EU
* Agreeable to utilize medically acceptable form of contraception
* Able to reconstitute and self-inject or have a designee

Exclusion Criteria:

* Withdrawn from study 0881A3-312-EU
* Abnormal hematology or chemistry profiles
* Clinically relevant medical conditions including: congestive heart failure, multiple sclerosis or other central demyelinating diseases, blood dyscrasias, cancer or serious infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety of etanercept in adults with ankylosing spondylitis who have completed study 0881A3-312-EU.

SECONDARY OUTCOMES:
To assess the long-term clinical efficacy of etanercept in these study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer